CLINICAL TRIAL: NCT06290024
Title: A Multi-center Clinical Longitudinal Study of Neuropathic Pain by Collecting Data on Patients' Brain Physiology and Cognitive Function
Brief Title: A Multi-center Clinical Longitudinal Study of Neuropathic Pain by Collecting Data
Status: Recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-23-013
Record Dates: First submitted 2023-12-26; First posted 2024-03-04 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with neuropathic pain: With prospective and longitudinal research design, patients with neuropathic pain that meet the entry/displacement standards will be included in the group and receive the routine diagnosis and treatment of the pain department. At the same time, the patients admitted to the group will be clinical observation and studied. After the diagnosis and treatment, follow-up will be carried out until 3 months after joining the group.
  Interventions: Device: A multi-center clinical longitudinal study of neuropathic pain by collecting data on patients' brain physiology and cognitive function

INTERVENTIONS:
Device: A multi-center clinical longitudinal study of neuropathic pain by collecting data on patients' brain physiology and cognitive function — Using the use of pain visual analog scale (VAS), digital pain grading method (NRS), neuropathic pain assessment scale (DN4), sleep quality (Pittsburgh sleep quality index, Ascens insomnia scale), social support assessment scale (SSQ), Montreal cognitive assessment scale (MoCA), Barrett impulse scale (BIS), anxiety and depression score (GAD-7, PHQ-9), emotional tasks, cognitive function (N-back, time perception, delay-discount), electroencephalogram (EEG), near-infrared brain function imaging (fNIRS) and other indicators to study the dynamic changes of various factors in the process of acute pain.

SUMMARY:
A multi-center clinical longitudinal study of neuropathic pain by collecting data on patients' brain physiology and cognitive function

DETAILED DESCRIPTION:
Using the use of pain visual analog scale (VAS), digital pain grading method (NRS), neuropathic pain assessment scale (DN4), sleep quality (Pittsburgh sleep quality index, Ascens insomnia scale), social support assessment scale (SSQ), Montreal cognitive assessment scale (MoCA), Barrett impulse scale (BIS), anxiety and depression score (GAD-7, PHQ-9), emotional tasks, cognitive function (N-back, time perception, delay-discount), electroencephalogram (EEG), near-infrared brain function imaging (fNIRS) and other indicators to study the dynamic changes of various factors in the process of acute pain.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participated in the study and signed an informed consent form;
2. The age is between 18 years old (inclusive) and 85 years old (inclusive), regardless of gender;
3. Body mass index (BMI) ≤ 45;
4. Clinically clearly diagnosed neuropathological pain (pain VAS score ≥4 or above);
5. Did not participate in the drug/medical device test within 3 months before the test;

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients who are in poor condition and cannot objectively describe their symptoms or complete the questionnaire score;
  2. People with severe mental system, respiratory system, cardiovascular system diseases, liver and kidney insufficiency, malignant tumors;
  3. Lactation, pregnant women, or subjects with pregnancy plans within 1 month after the trial (including male subjects);
  4. People with allergic diseases and allergic constitution;
  5. People with infected or damaged skin at the EEG collection site;
  6. Have a history of drug abuse or drug addiction;
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale/Score（VAS） | 1 month
  VAS pain score criteria ((0-10 points) 0 Points: painless; 3 points below: have a slight pain, can tolerate; 4 points- -6 points: patients with pain and affect sleep, and can still tolerate; 7 points-10 points: the patient has gradually intense pain, the pain is unbearable, affect appetite, affect sleep.
digital pain grading method (NRS) | 1 month
  Score ranged from 1 to 5, and the higher the score, the more it suggested the possibility of neuropathic pain. Clinically, when patients score ID Pain 3, neuropathic pain-related treatment options will be considered.
neuropathic pain assessment scale (DN4) | 1 month
  Each assessment item was assigned 1 point for "yes" and 0 point for "no". The total score of DN4 is 0 to 10, and neuropathic pain when the total score is greater than or equal to 4.
sleep quality (Pittsburgh sleep quality index, Ascens insomnia scale) | 1 month
  The PSQI was used to assess the sleep quality of the participants in the last 1 month. It consists of 19 self-assessment entries and 5 items, among which the 19th self-assessment entry and 5 items do not participate in the scoring. Only the 18 self-assessment entries participating in the scoring are introduced here (see the attached questionnaire for details). The 18 items formed 7 components, and each component was scored according to 0-3 levels. The cumulative score of PSQI total score ranged from 0 to 2 l. The higher the score, the worse the sleep quality.
EEG | 1 month
  To study the dynamic change of EEG wavelength during the progression from acute pain to chronic pain，four basic waveforms, α, β, θ, δ wave, were collected。
Barrett impulse scale (BIS) | 1 month
  The subject's feeling, reaction and degree of recognition are regarded as evaluation indicators, and the five-point scale classification method is adopted. Action impulse is scored positively, and unplanned impulse and cognitive impulse are scored in reverse. The standard is: "1" means never or almost never; "2" means occasional; "3" means often; "4" means always or almost always.
(Generalized Anxiety Disorder,GAD-7) | 1 month
  Each entry is 0 to 3 points, the total score is the score of the 7 items, the total score ranges from 0 to 21 points A 0-4 score is found without a GAD And 5-9 points for mild GAD And 10 - 14 points for moderate GAD 15 - 21 for severe GAD
(Patient Health Questionnaire-9 | 1 month
  Calculate the total score 0-4 points: no depression (take care of yourself) 5-9: possible mild depression (consult a psychologist or medical worker recommended) 10-14 points: There may be moderate depression (preferably consult a psychologist or psychological medicine worker) 15-19: possible moderate to severe depression (consult a psychiatrist or psychiatrist) 20-27: possible severe depression (be sure to see a psychologist or psychiatrist) Core project points Item 1, item 4, item 9, any question score> 1 (select 2,3), need attention; item 1, item 4, representing the core symptoms of depression; Item 9 represents a self-injury mind.

SECONDARY OUTCOMES:
Montreal cognitive assessment scale (MoCA) | 1 month
  The Montreal Cognitive Assessment (Montreal Cognitive Assessment, MoCA) is a rating tool for rapid screening of cognitive abnormalities. It includes eight cognitive domains, including visual structure skills, executive function, memory, language, attention and concentration, calculation, abstract thinking and directional force. The total score of 30 and 26 were normal, with high sensitivity, covering important cognitive fields, short test time and suitable for clinical use.
ocial support assessment scale (SSQ) | 1 month
  Each group of questions asked (A) how satisfied you are with the number of people who help or support you in your life, and (B) how satisfied you are with the way they / they help you.1= very dissatisfied, and 6= very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: ke na ma, phd, Study Chair — studay chair
Locations (1):
- Ke Ma, Shanghai, Yangpu, China

IPD SHARING:
Plan to Share IPD: Undecided